CLINICAL TRIAL: NCT01567618
Title: A Phase II Trial Evaluating Biweekly Docetaxel and DeGramont Regimen in First-Line Treatment of Unresectable or Metastatic Gastric Adenocarcinoma (DaeMon)
Brief Title: Dose-dense Biweekly Docetaxel Combined With 5-fluorouracil as First-line Treatment in Advanced Gastric Cancer
Acronym: DaeMon
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jian Xiao, Principal Investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAHMO-04
Record Dates: First submitted 2012-03-27; First posted 2012-03-30 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Gastric Adenocarcinoma
Keywords: Docetaxel; Fluorouracil; First line therapy; Gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Docetaxel — Docetaxel 50mg/m2 iv drip, repeat every two weeks;
  Efficacy will be evaluated every three cycles.
Drug: Fluorouracil — Fluorouracil 400mg/m2 iv D1; Fluorouracil 2400mg/m2 civ 46 hours; repeat fortnightly and evaluate every two cycles

SUMMARY:
This is an open-label, phase II study to evaluate the efficacy and safety of biweekly docetaxel and DeGramont regimen on unresectable gastric adenocarcinoma in the first-line therapy.

DETAILED DESCRIPTION:
Primary endpoint: Overall Response Rate

Secondary endpoint: Time to progression, overall survival, safety data

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Patients with histologically or cytologically confirmed unresectable gastric adenocarcinoma whose ECOG performance status are 0-2
* Presence of measurable disease by radiographic study (including CT or MRI scan, or chest x-ray) or physical examination
* At least 3 weeks since last major surgery
* At least 12 months since last adjuvant chemotherapy
* At least 6 weeks since prior radiotherapy providing that the extent and site of radiotherapy fields are such that marked bone marrow suppression is NOT expected
* Patients who have received palliative radiotherapy must have recovered from any reversible toxic effects e.g. nausea and vomiting caused by radiation of fields
* Patients with reproductive potential must use effective BC;
* Required Screening Laboratory Criteria:

Hemoglobin 90g/L WBC 3.5 x 109/L Neutrophils 1.5 x 109/L Platelets 100 x 109/L Creatinine 133 umol/L and creatinine clearance 60 mL/min

* A probable life expectancy of at least 6 months;

Exclusion Criteria:

* Brain metastases
* Female of childbearing potential, pregnancy test is positive
* Concomitant malignancies or previous malignancies other than gastric cancer within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or low grade prostate cancer
* Active infection
* Concurrent severe medical problems unrelated to the malignancy, which would significantly limit full compliance with the study or expose the patient to extreme risk
* Sexually active patients refusing to practice adequate contraception; Patients with conditions which might affect absorption of an oral drug (for example intermittent obstruction) unless discussed and agreed with principal investigator
* History of grade 3 or 4 toxicity to fluoropyrimidines

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-03; Primary Completion 2013-09 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate according to RECIST 1.1 | One Year

SECONDARY OUTCOMES:
Time to progression | One year
Overall survival | One year
Incidence of grade 3 or 4 toxicity | One year
  The criteria to grade the toxicity is NCI CTC 3.0

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China